CLINICAL TRIAL: NCT03427801
Title: Effect of Erythropoiesis-Stimulating Agent Therapy in Patients Receiving Palliative Care of Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chow Kai Ming, Dr, Chinese University of Hong Kong
Other Study IDs: CREC2017.147
Record Dates: First submitted 2018-02-03; First posted 2018-02-09 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: erythropoiesis-stimulating agent
MeSH Terms: interventions — Hematinics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treatment Group: Chronic kidney disease patient receiving palliative care and erythropoiesis-stimulating agent
  Interventions: Drug: Erythropoiesis-Stimulating Agent
- Control Group: Chronic kidney disease patient receiving palliative care without erythropoiesis-stimulating agent

INTERVENTIONS:
Drug: Erythropoiesis-Stimulating Agent — erythropoiesis-stimulating agent: Mircera or Darbepoietin
  Groups: Treatment Group

SUMMARY:
An observational study to evaluate the effect of erythropoiesis-stimulating agents in treating anaemia of renal disease among adult patients receive palliative care instead of dialysis.

DETAILED DESCRIPTION:
Erythropoiesis-stimulating agent (ESA) has been commonly used to manage patients with end-stage renal disease receiving dialysis. The effects of ESA, however, are unclear. This study compares the result of erythropoiesis-stimulating agent (ESA) versus supportive care for chronic kidney disease patients receiving palliative care. The investigators design a retrospective observational study to evaluate the effect of erythropoiesis-stimulating agents in treating anaemia of renal disease among adult patients receive palliative care instead of dialysis. The primary objective is to assess whether ESA can reduce the transfusion burden and hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years and older, who opted for ESA treatment during palliative renal care for > 360 days between January 1, 2014 and December 31, 2016

Exclusion Criteria:

* patients who had dialysis or kidney transplant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with stage 4 to 5 chronic kidney disease undergoing palliative care pathway
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
number of red cell transfusion | one year
days of hospitalisation | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No